CLINICAL TRIAL: NCT01433133
Title: Phase I-II, Open Label, Uncontrolled, Dose Escalation Study of the Safety, Tolerability and Biologic Activity of the INFRADURE Biopump Secreting Sustained Interferon Alpha-2b (IFNα), in Combination With Oral Ribavirin for Genotype 3 Newly Diagnosed Hepatitis C Patients
Brief Title: Safety and Biological Activity of InfraDure Biopump Secreting Sustained Interferon in HCV Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company strategic decision
Sponsor: Medgenics Medical Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-002-02
Record Dates: First submitted 2011-09-05; First posted 2011-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): • Genotype 3 chronic HCV with detectable serum HCV RNA
  Interventions: Biological: implantation

INTERVENTIONS:
Biological: implantation — subcutaneous implantation of autologous dermis implant treated ex vivo with genetic vector carrying the gene for interferon alfa 2b

SUMMARY:
This will be a Phase I-II, open-label, single center, uncontrolled, dose-escalation study. The trial will be conducted in Israel at the Tel Aviv Sourasky Medical Center.

All subjects will receive autologous InfraDure Biopump (micro-organ of dermis processed ex vivo transduced with genetic construct containing the gene for interferon)tissue implants intended to provide sustained production and delivery of therapeutic levels of INF for up to twenty four (24) weeks following INFRADURE Biopump implantation. Follow up will continue for a total of two years post INFRADURE Biopump implantation

DETAILED DESCRIPTION:
Medgenics Inc. and Medgenics Medical Israel Ltd. are developing INFRADURE, an autologous dermal biopump capable of sustained secretion of therapeutic INF in the body, using a small tissue explant from the patient's own skin. The INFRADURE biopump is produced from a micro-organ (MO), typically measuring 30 mm in length and 1.5-2.5 mm diameter, which is harvested directly from the patient's dermis under local anesthesia. The micro-organ can be viably maintained ex-vivo for extended periods of time under standard culture conditions. INFRADURE Biopumps, produced by ex vivo transduction of MOs with Helper Dependent Adenoviral INF vectors (HDAd-INF), express and secrete INF. INFRADURE Biopump is monitored ex vivo prior to re-implantation, to attain true INF dosing. The INFRADURE Biopump is subsequently implanted subcutaneously back to the patient in order to provide continuous delivery of a known amount of INF. Each implanted autologous INFRADURE Biopump remains localized under the skin, and is accessible, so that if necessary, it can be removed or ablated at any time. The entire process from harvest to implantation requires 10-14 days

ELIGIBILITY:
Inclusion Criteria:

* Signed patient consent form
* Genotype 3 chronic HCV with detectable HCV RNA
* No previous treatment for HCV infection
* Hepatitis B and human immunodeficiency virus negative at screening visit
* Able and willing to follow contraception requirements
* Screening laboratory values, test, and physical exam within acceptable ranges

Exclusion Criteria:

* Current enrollment in another investigational device or drug study
* Anticipated inability to complete all clinic visits and comply with study procedures
* History of, or any current medical condition, which could impact the safety of the subject during the study
* Autoimmune hepatitis, suspected hepatocellular carcinoma, decompensated liver disease, or other known liver disease other than HCV
* Alcoholism or substance abuse with <6 documented months of sobriety
* Known allergy or sensitivity to interferons or ribavirin
* Any other condition that, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Viral Load: incidence of sustained virologic response (SVR) | 24 weeks
  Viral load to be measured along the study expecting notable decrease in the viral load by week 24 post intervention

SECONDARY OUTCOMES:
Rapid virologic response (RVR) | Time Frame-Study Week 4
Early virologic response (EVR) | Time Frame-Study week 12
End-of-treatment response (EOT) | Time Frame-Study week 48, 104
Rapid virologic response (RVR) | Evaluation after 4 weeks from treatment day 0

IPD SHARING:
Plan to Share IPD: No